CLINICAL TRIAL: NCT04468867
Title: Role of ABUS as an Alternative to Breast MRI in Assessing Response to Neoadjuvant Chemotherapy
Acronym: RABUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD19/121361
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (Experimental)
  Interventions: Diagnostic Test: Automated whole breast ultrasound; Diagnostic Test: Breast MRI

INTERVENTIONS:
Diagnostic Test: Automated whole breast ultrasound — This will be performed by a band 6 radiographer and will be done at baseline, post 2 cycles of chemotherapy and end of treatment chemotherapy
Diagnostic Test: Breast MRI — This will be performed by band 6 or 7 radiographer with MRI training

SUMMARY:
Some women who have been diagnosed with a breast cancer will require chemotherapy as part of their treatment. The chemotherapy can be given before breast surgery - neoadjuvant chemotherapy or after breast surgery - adjuvant chemotherapy. Whether chemotherapy is given before or after does not affect the clinical outcomes for the woman - ie there is no disadvantage to the woman. Due to the fact that giving chemotherapy before has no disadvantages, many of the oncologists like to give the chemotherapy before because they can see if the breast cancer is responding. They are able to do this by using imaging. The best imaging test is breast MRI. Ultrasound can be used but studies have shown that it is not as good. However, whole breast ultrasound (ABUS) provides 3 dimensional information similar to breast MRI and the purpose of our study is to see if ABUS performs similar to breast MRI in being able to see if a tumour is responding to the chemotherapy. The breast MRI requires women to lie facing down and takes about 20mins. It involves an injection of contrast called gadolinium via a cannula. ABUS involves scanning the whole breast with the patient lying on their back and takes 10mins. There is no injection of contrast. MRI is an expensive test and often there is limited access to the scanner and so patients may have to wait for an appointment. ABUS because it is an automated process for obtaining the images can be performed in the breast unit in a timely manner without the issue of competing demands. All women who agree to take part in the study will have both the breast MRI - standard or care and the ABUS.

ELIGIBILITY:
Inclusion Criteria:

1. All female participants eligible for neoadjuvant chemotherapy and planning surgical treatment
2. Able to give informed consent

Exclusion Criteria:

1. All female particpants having neoadjuvant chemotherapy as palliative treatment with no surgery planned
2. Unable to provide informed consent
3. Unable to have breast MRI scan due to clautrophobia or allergy to gadolineum

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumour size | 20 mins
  Response will be assessed using RECIST criteria. Longest diameter response was scored based on the RECIST guidelines (PD>20% increase, SD<20% increase to<30% decrease, PR>30% decrease in longest diameter and CR if no tumour is visible).

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom